CLINICAL TRIAL: NCT00281541
Title: A Phase II, Multicenter, Open-Label Study of YM155 in Subjects With Unresectable Stage III or Metastatic (Stage IV) Melanoma
Brief Title: A Study for the Treatment of Unresectable Stage III or Metastatic Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-008
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
Keywords: Treatment Efficacy; Treatment Effectiveness; Disease Management; Treatment; Safety; Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — sepantronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YM155

SUMMARY:
A study with YM155 for the treatment of unresectable stage III or metastatic stage IV melanoma.

DETAILED DESCRIPTION:
A phase II, multicenter, open-label study in subjects with unresectable Stage III or metastatic (Stage IV) Melanoma to evaluate the efficacy and safety of YM155

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable stage III or IV malignant melanoma
* Life expectancy >12 weeks

Exclusion Criteria:

* History of other malignancy in the last 5 years
* Major surgery within the past 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2005-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | 6 cycles

SECONDARY OUTCOMES:
Duration of response | 6 cycles

CONTACTS AND LOCATIONS:
Overall Officials: D. Buell, MD, Study Director — Astellas Pharma US, Inc.
Locations (9):
- United States (9):
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Montclair, New Jersey
  - Winston-Salem, North Carolina
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah